CLINICAL TRIAL: NCT05456659
Title: Renal Replacement Therapy in Neonates : a Retrospective Monocentric Cohort Study
Brief Title: Renal Replacement Therapy in Neonates
Acronym: Neo-Renal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8615
Record Dates: First submitted 2022-04-27; First posted 2022-07-13 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-04

CONDITIONS: Renal Failure
Keywords: Neonatal; Dialysis; Extra-renal purification; Neonatal resuscitation
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The circumstances for setting up dialysis in the neonatal period are multiple: congenital anomaly of the kidney and urinary tract (CAKUT), secondary acute renal failure whose etiologies are multiple (sepsis, hypovolemia, respiratory distress syndrome, neonatal asphyxia, Arterial or venous renal thrombosis, nephrotoxic drugs, etc.), metabolic diseases (mainly hyperammonemia and leucinosis) and post-operative management of heart disease: analysis of the characteristics of the patients in our study and comparison with existing epidemiological data in the literature.

The decision to set up dialysis in a newborn whose recovery of renal function is uncertain or in a context of acute multi-visceral failure is not always obvious and must be discussed carefully. multidisciplinary in connection with neonatologists, resuscitators and nephrologists as well as families with the consideration of the future quality of life of the child.

ELIGIBILITY:
Inclusion criteria:

* Minor under 28 days old
* Having benefited from a renal purification technique in the pediatric intensive care unit of the University Hospital of Strasbourg
* Holders of parental authority who do not object to the reuse of their child's data for scientific research purposes.

Exclusion criteria:

- Holders of parental authority who have expressed their opposition to the reuse of their child's data for scientific research purposes.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor under 28 days old, having benefited from a renal purification technique in the pediatric intensive care unit of the University Hospital of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-10-27 (Estimated); Study Completion 2022-10-27 (Estimated)

PRIMARY OUTCOMES:
Description of clinical characteristics of patients, survival and technical modalities of dialysis in children undergoing neonatal dialysis at the Strasbourg University Hospital | Files analysed retrospectively from January 01, 2010 to December 31, 2021 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France